CLINICAL TRIAL: NCT04647435
Title: National, Multicentre, Randomized, Double-blind, Triple-dummy Active-Controled Phase III Clinical Trial to Evaluate the Efficacy and Safety of APSCTC for the Treatment of Postsurgical Pain Due to Third Molar Extraction.
Brief Title: Efficacy and Safety of APSCTC for the Treatment of Postsurgical Pain Due to Third Molar Extraction
Acronym: CARLOTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apsen Farmaceutica S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APS001/2020
Record Dates: First submitted 2020-11-18; First posted 2020-12-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Postsurgical Pain; Third Molar Extraction
MeSH Terms: conditions — Pain, Postoperative | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- APSCTC (Experimental): Oral tablets every 6h for 3 days
  Interventions: Drug: APSCTC
- Toragesic® (Active Comparator): Oral tablets every 6h for 3 days
  Interventions: Drug: Toragesic®
- Tramal® (Active Comparator): Oral tablets every 6h for 3 days
  Interventions: Drug: Tramal®

INTERVENTIONS:
Drug: APSCTC — APSCTC + Toragesic® placebo + Tramal® placebo
  Arms: APSCTC
Drug: Toragesic® — APSCTC placebo + Toragesic® + Tramal® placebo
  Arms: Toragesic®
Drug: Tramal® — APSCTC placebo + Toragesic® placebo + Tramal®
  Arms: Tramal®

SUMMARY:
The purpose of this study is to evaluate the efficacy of APSCTC compared to two active drugs in acute pain relief.

ELIGIBILITY:
Main Inclusion Criteria:

* Males and Females aged 18 to 40 years;
* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants who require extraction of impacted mandibular third molar.

Main Exclusion Criteria:

* Known hypersensitivity to the formula components used during the clinical trial;
* Previous history of alcohol or drugs abuse diagnosed by DSM-V;
* Previous history of renal failure from moderate to severe;
* Women who are pregnant, lactating, or positive for β - hCG urine test.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

PRIMARY OUTCOMES:
At least 50% of maximum pain relief score (TOTPARmax) | Change from Baseline to 6 hours

SECONDARY OUTCOMES:
Adverse events incidence and classification | During treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Azidus Brasil Pesquisa Científica e Desenvolvimento Ltda., Valinhos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No